CLINICAL TRIAL: NCT06217458
Title: The Added Value of Contrast Enhanced Mammography (CEM) to Standard Mammography in Assessing the Extent of Ductal Carcinoma in Situ (DCIS)
Brief Title: The Added Value of Contrast Enhanced Mammography to Standard Mammography in Assessing the Extent of DCIS
Acronym: CEMinDCIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Center Rijeka (Other)
Responsible Party: Principal Investigator, Petra Valkovic Zujic, Head of Abdominal and Breast Division Department of Radiology, Clinical Hospital Center Rijeka
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: The added value of CEM
Record Dates: First submitted 2023-12-10; First posted 2024-01-22 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: DCIS; Breast Carcinoma in Situ; Calcification
Keywords: Ductal in situ carcinoma; Calcifications; Breast surgery; Screening; Contrast Enhanced Mammography
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Calcinosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Patients with mammographically newly detected ductal in situ carcinoma who undergo surgery at CHC Rijeka in 2024, 2025, and 2026 (consecutively), who agree to have a CEM performed prior to surgery as part of the diagnostic work-up in addition to standard mammography, and who agree to participate in the examination. Group number: 50 patients.
  Interventions: Diagnostic Test: Contrast Enhanced Mammography
- Historical Control (No Intervention): Patients diagnosed with ductal in situ carcinoma who underwent surgery at CHC Rijeka in the period from 2019 to 2024 and whose clinical data are available in the prospectively managed clinical registry for breast diseases at CHC Rijeka and in the Hospital Information System (IBIS). Group number: 50 patients.

INTERVENTIONS:
Diagnostic Test: Contrast Enhanced Mammography — The CEM performance protocol involves the intravenous administration of non-ionic, low-osmolarity iodinated contrast medium using an automatic syringe that delivers the required bolus of contrast medium at a dose of 1.5 ml/kg body weight at a rate of 3 ml/s without compressing the breast. After a two-minute pause, necessary to allow the breast parenchyma to absorb (stain) the contrast agent, the patient is positioned for the mammogram and the breast is compressed. First the symptomatic and then the non-symptomatic breast is imaged in two or a total of four standard projections: craniocaudal (CC) and oblique mediolateral (MLO) projections of the breast. The delayed CC and MLO projections of the symptomatic breast are taken within eight minutes of the start of the examination. The delayed mammograms are used to assess the dynamics of the contrast uptake of the lesion and are compared to the same parameters of the breast MRI. The time required to perform the CEM is 8-10 minutes.
  Other Names: CEM
  Arms: Interventional Group

SUMMARY:
The study hypothesis is that the rate of inadequate surgical margins after conservative breast surgery for DICS and the rate of reoperation (re-excision or/and mastectomy) is lower in the group of patients who underwent standard preoperative mammography and CEM to assess the extent of DICS, compared to the group of patients for whom the preoperative assessment of the extent of in situ breast cancer was not performed using one of the imaging techniques with contrast medium such as contrast mammography or magnetic resonance imaging.

DETAILED DESCRIPTION:
Ductal carcinoma in situ (DCIS) is the earliest form of malignant lesion in the breast, which in most cases is diagnosed by mammography screening, usually in the form of asymptomatic calcifications. The question of whether DCIS is a true malignancy of the breast, which pathological criteria are used for diagnosing and classifying DCIS, but also the questions of the nature of the disease and its overtreatment are controversial. Surgery is still the primary treatment of DCIS, and the status of the surgical margins is of paramount importance. Compared to invasive ductal carcinoma, the re-excision rate in DCIS is relatively high (30-40%), probably because the change is not palpable. Segmental distribution, with areas affected by the disease that are not calcified and therefore not detected, and stricter guidelines for appropriate surgical margins may also contribute to the re-excision rate. Because the diagnosis of DCIS is closely associated with mammographic detection of pathologic calcifications, it was assumed that magnetic resonance (MR) imaging would provide little or no value for their detection and visualization. However, a study conducted by Kuhl et al. showed that breast MRI has a significantly higher sensitivity than mammography in detecting DCIS. In addition, subsequent studies have shown that MRI is more accurate than mammography in assessing the distribution of DCIS. In recent years, mammography with an iodine contrast agent, known as contrast mammography (CEM), has been introduced, which, like MRI, is based on the evaluation of tumor angiogenesis. It is important to emphasize that the sensitivity of CEM in detecting malignant lesions corresponds to the sensitivity of MR. CEM has several advantages over breast MRI, the most important of which are the availability and the shorter imaging time, as well as the shorter time required to analyze the mammogram and read the findings. Numerous studies show that patients tolerate CEM better than MRI.

The study hypothesis is that the rate of inadequate surgical margins after conservative breast surgery for DICS and the rate of reoperation (re-excision or/and mastectomy) is lower in the group of patients who underwent standard preoperative mammography and CEM to assess the extent of DICS, compared to the group of patients for whom the preoperative assessment of the extent of in situ breast cancer was not performed using one of the imaging techniques with contrast medium, such as contrast mammography or magnetic resonance imaging. The interventional cohort involves 50 consecutive patients with newly diagnosed DCIS who will undergo surgery at CHC Rijeka in 2024, 2025, and 2026 and who agree to have a CEM performed before surgery as part of the diagnostic work-up in addition to standard mammography and who agree to participate in the trial. Patients diagnosed with ductal in situ carcinoma who underwent surgery at CHC Rijeka in the period from 2019 to 2024 and whose clinical data are available in the prospectively managed clinical register for breast diseases at CHC Rijeka and the Integrated Hospital Informatics System (IBIS), are included in the second (control) cohort.

Two clinical radiology specialists with experience in breast radiology will evaluate the morphologic and functional features of standard MMG and CEM by consensus, and assess the extent of disease using the BI-RADS lexicon for imaging with contrast mammography. Demographic and imaging data (morphological and functional characteristics on CME such as background parenchymal enhancement, presence/absence of a lesion, location of the lesion in breast quadrant, type of lesion, size of the lesion in mm and BI-RADS category are analyzed for each lesion) will be recorded. Only one lesion per breast is considered, and if multiple lesions are visible, the overall diameter of the suspicious area will be considered. The above parameters are compared with the grade of the DCIS tumor, i. e. the morphological and functional characteristics of G1 and G2 lesions compared to G3 lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathohistological diagnosis of ductal in situ carcinoma based on samples obtained by vacuum-assisted breast biopsy (VABB) or ultrasound-guided breast biopsy (CNB)
* Presented at the meeting of the multidisciplinary breast team of the Clinical Hospital Center in Rijeka
* Patients who underwent surgery at CHC Rijeka and whose pathohistological diagnosis in the final PH report was pure DCIS or microinvasive breast cancer (DCIS with microinvasion)
* Patients who agree to participate in the study

Exclusion Criteria:

* Patients with contraindications for CEM: renal insufficiency (which is ruled out by presenting creatinine and/or eGFR results), iodine allergy, pregnancy/lactation, hyperthyroidism
* Patients who have undergone a preoperative breast MRI
* Patients who have both DCIS and invasive carcinoma in the preoperative PH report or the final PH report of the surgical material, with the exception of foci with microinvasion (< 1 mm).
* Patients with ipsilateral DCIS recurrence or with previous ipsilateral breast surgery for invasive cancer.
* Patients/subjects whose CEMs do not correspond to the diagnostic interpretation for technical reasons are excluded from the study: insufficient positioning, contrast agent extravasation, failed subtraction
* Patients under 18 years of age

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of true positive CEMs in the Interventional group | 3 years
  Number of patients in whom the estimated size of DCIS (longest diameter in mm) is larger on CEM than on MMG and in whom the actual size in PH report is greater than the size on estimated on MMG
Number of false positive CEMs in the Interventional Group | 3 years
  Number of patients in whom the estimated size of DCIS (longest diameter in mm) on CEM is larger than on MMG, but the size in the PH report correlates better with the size estimated on MMG
Number of true negative CEMs in the Interventional Group | 3 years
  Number of patients with no difference in the radiological assessment of the size of DCIS (longest diameter in mm), and in whom the size in the PH report correlates with the size on MMG
Number of false negative CEMs in the Interventional Group | 3 years
  Number of patients with no difference in the radiological assessment of the size of DCIS (longest diameter in mm is similar on CEM and MMG), but in whom the size in the PH report is greater than the size on MMG and CEM
True positive rate of CEM vs. MMG (Sensitivity) | 3 years
  True positive rate = Number of true positive / (Number of true positive + Number of false negative)
True negative rate of CEM vs. MMG (Specificity) | 3 years
  True negative rate = Number of true negative / (Number of true negative + Number of false positive)
False positive rate of CEM vs. MMG (overestimation) | 3 years
  False positive rate = Number of false positive / (Number of false positive + Number of true negative)
False negative rate of CEM vs. MMG (underestimation) | 3 years
  False negative rate= Number of false negative / (Number of false negative + Number of true positive)
Accuracy of CEM vs. MMG | 3 years
  Accuracy = (Number of true positive + Number of true negative) / (Number of true positive+ Number of false positive + Number of true negative + Number of false negative)
Inadequate surgical margins rate in the Interventional Group | 3 years
  Percentage of patients with inadequate surgical margins (<2mm)
Inadequate surgical margins rate in the Control Group | 3 years
  Percentage of patients with inadequate surgical margins (<2mm)
Re-operation rate in the Interventional Group | 3 years
  Percentage of repeated surgical procedures in breast
Re-operation rate in the Control Group | 3 years
  Percentage of repeated surgical procedures in breast
Mastectomy rate in the Interventional Group | 3 years
  Percentage of patients with mastectomy
Mastectomy rate in the Control Group | 3 years
  Percentage of patients with mastectomy

SECONDARY OUTCOMES:
Estimated percentage of breast resection volume based on CEM | 3 years
  Percentage of breast resection volume based on CEM findings according to the formula (4 x (radius of the lesion + 1 cm)3 ) : (radius of the breast 2 x projection of the breast)
Estimated percentage of breast resection volume based on MMG | 3 years
  Percentage of breast resection volume based on MMG findings according to the formula (4 x (radius of the lesion + 1 cm)3 ) : (radius of the breast 2 x projection of the breast)
Duration of complete preoperative diagnostic workup in the Intervention Group | 3 years
  Number of days between the date of the first clinical examination at CHC Rijeka (surgeon or radiologist) and the date of surgery
Duration of complete preoperative diagnostic workup in the Control Group | 3 years
  Number of days between the date of the first clinical examination at CHC Rijeka (surgeon or radiologist) and the date of surgery
Lesion extension of high-grade DCIS (G3) on CEM | 3 years
  Size of the lesion determined in millimetres.
Lesion extension of low-grade DCIS (G1-2) on CEM | 3 years
  Size of the lesion determined in millimetres.
Background parenchymal enhancement associated with high-grade DCIS (G3) on CEM | 3 years
  Background parenchymal enhancement (symmetric or asymmetric) is categorized as minimal, mild, moderate and marked.
Background parenchymal enhancement associated with low grade DCIS (G1-2) on CEM | 3 years
  Background parenchymal enhancement (symmetric or asymmetric) is categorized as minimal, mild, moderate and marked.
Distribution of NME associated with high-grade DCIS (G3) on CEM | 3 years
  Non-mass enhancement (NME) classified as: focal, linear, segmental, regional, multiple regions or diffuse.
Distribution of NME associated with low grade DCIS (G1-2) on CEM | 3 years
  Non-mass enhancement (NME) classified as: focal, linear, segmental, regional, multiple regions or diffuse.
Lesion conspicuity associated with high-grade DCIS (G3) on CEM | 3 years
  Lesion conspicuity (relative to background) is the degree of enhancement compared to background, described as low, moderate or high
Lesion conspicuity associated with low grade DCIS (G1-2) on CEM | 3 years
  Lesion conspicuity (relative to background) is the degree of enhancement compared to background, described as low, moderate or high
Morphologic features of mass lesion associated with high-grade DCIS (G3) on CEM | 3 years
  Mass lesions are defined by shape and margin: descriptors for mass shape and margin include oval, round, or irregular shape, with circumscribed or not circumscribed (irregular, spiculated) margin.
Morphologic features of mass lesion associated with low grade DCIS (G1-2) on CEM | 3 years
  Mass lesions are defined by shape and margin: descriptors for mass shape and margin include oval, round, or irregular shape, with circumscribed or not circumscribed (irregular, spiculated) margin.
Internal pattern of enhancement of mass lesion associated with high-grade DCIS (G3) on CEM | 3 years
  Internal pattern can be homogeneous, heterogeneous, or rim enhancement.
Internal pattern of enhancement of mass lesion associated low grade DCIS (G1-2) on CEM | 3 years
  Internal pattern can be homogeneous, heterogeneous, or rim enhancement.
Overall treatment cost in the Interventional Group | 3 years
  All costs related to diagnostic workup and related to surgical treatment will be evaluated for each patient (costs of the procedure, hospital days, readmission rate after the first treatment).
Overall treatment cost in the Control Group | 3 years
  All costs related to diagnostic workup and related to surgical treatment will be evaluated for each patient (costs of the procedure, hospital days, readmission rate after the first treatment).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital Centre Rijeka, Rijeka, Primorsko Goranska County, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Covington MF, Pizzitola VJ, Lorans R, Pockaj BA, Northfelt DW, Appleton CM, Patel BK. The Future of Contrast-Enhanced Mammography. AJR Am J Roentgenol. 2018 Feb;210(2):292-300. doi: 10.2214/AJR.17.18749. Epub 2017 Oct 24. PMID 29064748
- [Background] Covington MF. Contrast-Enhanced Mammography Implementation, Performance, and Use for Supplemental Breast Cancer Screening. Radiol Clin North Am. 2021 Jan;59(1):113-128. doi: 10.1016/j.rcl.2020.08.006. Epub 2020 Oct 29. PMID 33222993
- [Background] Kuhl CK, Strobel K, Bieling H, Wardelmann E, Kuhn W, Maass N, Schrading S. Impact of Preoperative Breast MR Imaging and MR-guided Surgery on Diagnosis and Surgical Outcome of Women with Invasive Breast Cancer with and without DCIS Component. Radiology. 2017 Sep;284(3):645-655. doi: 10.1148/radiol.2017161449. Epub 2017 Apr 26. PMID 28445683
- [Background] Sardanelli F, Trimboli RM, Houssami N, Gilbert FJ, Helbich TH, Alvarez Benito M, Balleyguier C, Bazzocchi M, Bult P, Calabrese M, Camps Herrero J, Cartia F, Cassano E, Clauser P, Cozzi A, de Andrade DA, de Lima Docema MF, Depretto C, Dominelli V, Forrai G, Girometti R, Harms SE, Hilborne S, Ienzi R, Lobbes MBI, Losio C, Mann RM, Montemezzi S, Obdeijn IM, Ozcan UA, Pediconi F, Pinker K, Preibsch H, Raya Povedano JL, Sacchetto D, Scaperrotta GP, Schiaffino S, Schlooz M, Szabo BK, Taylor DB, Ulus OS, Van Goethem M, Veltman J, Weigel S, Wenkel E, Zuiani C, Di Leo G. Magnetic resonance imaging before breast cancer surgery: results of an observational multicenter international prospective analysis (MIPA). Eur Radiol. 2022 Mar;32(3):1611-1623. doi: 10.1007/s00330-021-08240-x. Epub 2021 Oct 13. PMID 34643778
- [Result] Klaric K, Sribar A, Budisavljevic A, Labinac L, Valkovic Zujic P. Evaluation of Contrast-Enhanced Mammography and Development of Flowchart for BI-RADS Classification of Breast Lesions. Diagnostics (Basel). 2023 Jun 3;13(11):1958. doi: 10.3390/diagnostics13111958. PMID 37296810